CLINICAL TRIAL: NCT01442844
Title: Secondary Intention Wound Healing Versus Micrografting in Patients Undergoing Mohs Surgery
Acronym: MomelanMohs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study sponsor was acquired by a company that focuses on chronic wounds
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Momelan Technologies (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010p002614
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Impaired Wound Healing
Keywords: Mohs; Scalp

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micrografting (Active Comparator): Several small pieces of skin, each measuring 1.75 mm in diameter will be harvested from a normal pigmented area using a commercially available suction blister device. This will be attached to a sterile dressing that will be placed on the surgical wound.
  Interventions: Device: Micrografting
- No intervention (No Intervention): No intervention will be performed. Subject will receive dressings that are standard of care.

INTERVENTIONS:
Device: Micrografting — Several small pieces of skin, each measuring 1.75 mm in diameter will be harvested from a normal pigmented area using a commercially available suction blister device. This will be attached to a sterile dressing that will be placed on the surgical wound.
  Arms: Micrografting

SUMMARY:
This study evaluates a novel micrografting technique to see how it will influence the healing rate and cosmetic result of second intention wounds. The graft harvesting and micrografting process was designed by MoMelan Technologies The Epidermal Expansion System, which is composed of a commercially available Blister Generation Device and the Microblister Generation and Excision Device (MBGED), will generate an array of small microblisters and transfer the micrografts to a sterile dressing (Tegaderm™ - an FDA approved wound dressing) for application to the subject's surgical area. The investigators predict that applying expanded micrografts to wounds that otherwise would have healed by second intention alone will hasten healing and possible reduce scarring.

DETAILED DESCRIPTION:
Participants with a scalp wound s/p Mohs procedure will be randomized to a micrografting technique intervention or to no intervention/heal with secondary intention alone (control). Intervention consists of harvesting skin micrografts (1.75mm) from pigmented skin using the Microblister generation and excision device and transfer the micrografts to a sterile dressing for application to the participants scalp wound. Percent wound re-epithelialization will be compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Between 40-75 years old
2. Status post Mohs procedure on the scalp with a wound that would otherwise be allowed to heal by second intention
3. Superficial would-at deepest of 2.0 mm or to superficial fat, but not deep to muscle
4. Area is less then 6 cm2 (wound diameter less than 2cm)

Exclusion Criteria:

1. Female patients who are breastfeeding, pregnant, or planning to become pregnant
2. Abnormal bleeding observed during initial Mohs procedure that would suggest a higher risk of post-operative bleeding
3. Subjects currently on immunosuppressive medications, chemotherapy or a cytotoxic agent
4. Participation in another interventional study with potential exposure to an investigational drug within past 30 days or planned study entry within 90 days after study entrance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mgh Curtis, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Micrografting | No Intervention
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micrografting | No Intervention | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 74 | 66.5 [63 to 70] | 69 [63 to 74]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wound Re-epithelialization
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: percentage of wound re-epithelialization
Arm/Group | Micrografting | No Intervention
Number analyzed (Participants) | 1 | 2
percentage of wound re-epithelialization | 50 | 37.5 [25 to 50]

ADVERSE EVENTS:
Arm/Group | Micrografting | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No